CLINICAL TRIAL: NCT05575414
Title: Outcomes of Pregnant Barbadian Women With Obesity: A Case Controlled Prospective Study of Didactic Dietary Intervention Compared to a Standard Education Tool
Brief Title: Diet Versus Control Pregnant Barbadian Women Gestational Weight Gain Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of The West Indies (Other)
Responsible Party: Principal Investigator, Tonya Johnson, Doctor, The University of The West Indies
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Gestational Weight Gain Study
Record Dates: First submitted 2022-10-05; First posted 2022-10-12 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Obesity; Gestational Weight Gain; Obesity, Maternal
Keywords: Obesity; Gestational Weight Gain; Pregnancy; Afro-Caribbean; Barbadian; Barbados
MeSH Terms: conditions — Obesity; Gestational Weight Gain; Pregnancy in Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Didactic Sessions (Experimental): Women will receive online nutrition education by a registered dietitian, in addition to the same standard patient education tool as the other arm.
  Interventions: Behavioral: Didactic dietary sessions; Behavioral: Education Tool
- Education Tool (Experimental): Women will receive a standard patient education tool in the form of a leaflet.
  Interventions: Behavioral: Education Tool

INTERVENTIONS:
Behavioral: Didactic dietary sessions — Three one-hour online nutrition group classes will be scheduled at 17, 21 and 29 weeks gestation (± 1 week). Nutrient dense foods and beverages and limiting the intake of added sugars, sodium and saturated fat will be encouraged, as well as reading the nutrition facts label, individual goal setting and self-monitoring. Physician recommended physical activity will be encouraged. Food and beverage intake data will be measured by 24-hour dietary recalls collected on three non-consecutive days. Data will be collected by telephone interview by a registered dietitian or dietary technician on four separate occasions: 16, 20 and 28 weeks gestation (± 1 week) and 36 weeks of gestation. Details on portions consumed will be estimated using standard measuring cups and household utensils. Nutrient intake will be generated using Vision Software Nutrient Analysis Software and the United States Department of Agriculture Food Composition Database, Food Data Central.
  Arms: Didactic Sessions
Behavioral: Education Tool — The standard patient education tool will take the form of a leaflet which will include 1. A definition of body mass index 2. A list of measures to be taken to limit weight gain in pregnancy. 3. A description of the major nutrients required in pregnancy (folate, iron, calcium, vitamin D and protein). and 4.A description of the six food groups with recommendations for the number of servings per day.

SUMMARY:
The researcher will study a group of pregnant Barbadians with BMI at booking of greater than or equal to 35. All of the women will be given leaflets telling them about healthy diets in pregnancy and how to limit weight gain. Half of the women will be sent to the dietitian for small group classes on diet and how to limit weight gain. The two groups of women will be compared to see which group gains more weight and which group has more complications during the pregnancy.

DETAILED DESCRIPTION:
More than 2100 pregnant women per annum deliver their babies at the Queen Elizabeth Hospital, the lone publicly-funded hospital providing secondary and tertiary-level obstetric care in Barbados. Routinely recorded data do not capture whether patients are overweight or obese. Thus, the prevalence of obesity is not known amongst this population. Additionally, these women are not routinely referred for dietician services, and thus the impact of dietician intervention is not known. The aim of this research is to determine whether a dietitian-led intervention could lead to decreased gestational weight gain and less incidence of foetal macrosomia in a sample of Barbadian women, with class II obesity, attending a public antenatal clinic. Prior studies examining gestational weight gain, found no statistically significance between groups when a BMI of 30 was used. It is hoped that by using a group with higher obesity a larger difference will be seen with the intervention. Participants with body mass index greater than 35kg/m^2 who meet the eligibility criteria will be selected from one of five antenatal clinics at the Queen Elizabeth Hospital on the island of Barbados. They will be randomised to either receive didactic dietary sessions or a standard education tool. Mean weight change will be compared amongst the two groups after delivery to determine if there was a decrease in gestational weight gain amongst the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Woman over 18 years old
* Live singleton pregnancy
* BMI of greater than or equal to 35kg/m^2
* Registered patient of the Queen Elizabeth Hospital Antenatal Clinic

Exclusion Criteria:

* Presence of gestational diabetes or chronic diabetes mellitus,
* Have had bariatric surgery
* Do not speak english
* Pregnancy with a multiple gestation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Mean change in gestational weight in kilograms in each arm of the trial | From enrolment until delivery
  Weight at or before delivery minus weight at enrolment

SECONDARY OUTCOMES:
Mean neonatal birth weight in grams in each arm of the trial | Within one hour of birth
  Weight of the neonate at birth
Incidence of pregnancy induced hypertension in each arm of the trial | Beyond 20 weeks gestation and prior to delivery
  New hypertension presenting after 20 weeks of pregnancy without significant proteinuria
Incidence of gestational diabetes in each arm of the trial | Beyond 20 weeks gestation and prior to delivery
  Defined using the National Diabetes Data Group (NDDG) criteria, which uses fasting, 1-hour, 2-hour, and 3-hour plasma glucose levels of 5.8mmol/L, 10.6mmol/L, 9.2mmol/L and 8.1mmol/L respectively diagnosed after 20 weeks gestation
Incidence of primary post partum haemorrhage in each arm of the trial | Within 24 hours of delivery
  The loss of 500 milliliters or more of blood from the genital tract within 24 hours of the birth of a baby. Postpartum haemorrhage will be further subclassified as minor (blood loss 500-1000 ml) or major (blood loss more than 1000 ml)27. Major postpartum haemorrhage will also be subdivided into moderate (1001-2000 ml) and severe (more than 2000 ml).
Incidence of low one minute APGAR score in each arm of the trial | After one minute of birth
  Defined as a score less than seven

OTHER OUTCOMES:
Rates of the various modes of delivery | At time of delivery
  A qualitative variable described as vaginal delivery, assisted vaginal delivery or caesarean section and obtained from the patient's labour record
Rates of Augmentation or Induction of labour | At the time of delivery
  Augmentation of labour. Induction of labour
Rates of preterm birth | From enrolment until delivery
  Birth before 37 completed weeks of pregnancy
Rates of admission to Neonatal Intensive Care Unit | From birth to one week of life
  A qualitative variable described as admitted or not admitted to the neonatal intensive care unit and obtained from the participant's infant medical record
Rates of the presence of foetal malformation | From enrolment until delivery
  A qualitative variable described as malformation present or not present and obtained form the participant's infant medical record
Rates of foetal death | From enrolment until delivery
  A qualitative variable described as foetus dead or alive and obtained from the medical record of the participant or the medical record of the participant's infant.

CONTACTS AND LOCATIONS:
Overall Officials: Damian AJ Best, DM MRCOG MSc, Study Director — University of the West Indies Cave hill Campus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Satpathy HK, Fleming A, Frey D, Barsoom M, Satpathy C, Khandalavala J. Maternal obesity and pregnancy. Postgrad Med. 2008 Sep 15;120(3):E01-9. doi: 10.3810/pgm.2008.09.1920. PMID 18824817
- [Background] Chu SY, Callaghan WM, Kim SY, Schmid CH, Lau J, England LJ, Dietz PM. Maternal obesity and risk of gestational diabetes mellitus. Diabetes Care. 2007 Aug;30(8):2070-6. doi: 10.2337/dc06-2559a. Epub 2007 Apr 6. PMID 17416786
- [Background] Yu Z, Han S, Zhu J, Sun X, Ji C, Guo X. Pre-pregnancy body mass index in relation to infant birth weight and offspring overweight/obesity: a systematic review and meta-analysis. PLoS One. 2013 Apr 16;8(4):e61627. doi: 10.1371/journal.pone.0061627. Print 2013. PMID 23613888
- [Background] Marchi J, Berg M, Dencker A, Olander EK, Begley C. Risks associated with obesity in pregnancy, for the mother and baby: a systematic review of reviews. Obes Rev. 2015 Aug;16(8):621-38. doi: 10.1111/obr.12288. Epub 2015 May 28. PMID 26016557
- [Background] Aune D, Saugstad OD, Henriksen T, Tonstad S. Maternal body mass index and the risk of fetal death, stillbirth, and infant death: a systematic review and meta-analysis. JAMA. 2014 Apr 16;311(15):1536-46. doi: 10.1001/jama.2014.2269. PMID 24737366
- [Background] Wolff S, Legarth J, Vangsgaard K, Toubro S, Astrup A. A randomized trial of the effects of dietary counseling on gestational weight gain and glucose metabolism in obese pregnant women. Int J Obes (Lond). 2008 Mar;32(3):495-501. doi: 10.1038/sj.ijo.0803710. Epub 2008 Jan 29. PMID 18227847
- [Background] Vinter CA, Jensen DM, Ovesen P, Beck-Nielsen H, Jorgensen JS. The LiP (Lifestyle in Pregnancy) study: a randomized controlled trial of lifestyle intervention in 360 obese pregnant women. Diabetes Care. 2011 Dec;34(12):2502-7. doi: 10.2337/dc11-1150. Epub 2011 Oct 4. PMID 21972411
- [Background] Lima Ferreira J, Voss G, Doria M, Sa Couto A, Principe RM. Benefit of insufficient gestational weight gain in obese women with gestational diabetes mellitus: A multicenter study in Portugal. Diabetes Metab Syndr. 2021 Jan-Feb;15(1):419-424. doi: 10.1016/j.dsx.2021.01.020. Epub 2021 Feb 8. PMID 33582580
- [Background] Olander EK, Hill B, Skouteris H. Healthcare Professional Training Regarding Gestational Weight Gain: Recommendations and Future Directions. Curr Obes Rep. 2021 Jun;10(2):116-124. doi: 10.1007/s13679-021-00429-x. Epub 2021 Feb 20. PMID 33609271
- [Background] Poston L, Bell R, Croker H, Flynn AC, Godfrey KM, Goff L, Hayes L, Khazaezadeh N, Nelson SM, Oteng-Ntim E, Pasupathy D, Patel N, Robson SC, Sandall J, Sanders TA, Sattar N, Seed PT, Wardle J, Whitworth MK, Briley AL; UPBEAT Trial Consortium. Effect of a behavioural intervention in obese pregnant women (the UPBEAT study): a multicentre, randomised controlled trial. Lancet Diabetes Endocrinol. 2015 Oct;3(10):767-77. doi: 10.1016/S2213-8587(15)00227-2. Epub 2015 Jul 9. PMID 26165396
- [Background] Institute of Medicine (US) and National Research Council (US) Committee to Reexamine IOM Pregnancy Weight Guidelines; Rasmussen KM, Yaktine AL, editors. Weight Gain During Pregnancy: Reexamining the Guidelines. Washington (DC): National Academies Press (US); 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK32813/ PMID 20669500